CLINICAL TRIAL: NCT02572622
Title: Lumbal Disk Herniasyonunda Farklı Tedavi Yöntemlerinin Karşılaştırılması
Brief Title: Comparison of Different Treatment Methods in Lumbal Disc Herniation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, research assistant Aynur Demirel, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HacettepeUN
Record Dates: First submitted 2015-07-15; First posted 2015-10-09 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Lumbar Disc Herniation
Keywords: exercise; deep friction massage; spinal decompression; non-surgical spinal decompression
MeSH Terms: conditions — Intervertebral Disc Displacement; Motor Activity | interventions — Electric Stimulation Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- spinal decompression group (Experimental): only 15 sessions of spinal decompression therapy were applied.
  Interventions: Other: non -surgical spinal decompression therapy
- combine group (Experimental): 10 patients participated in this group. for two weeks electrotherapy, deep friction massage and traction and last two weeks electrotherapy and exercise totally 15 session of treatment were applied.
  Interventions: Other: non -surgical spinal decompression therapy; Other: deep friction massage,; Other: electrotherapy; Other: exercise
- exercise group (Experimental): 10 patients participated in this group. for two weeks electrotherapy, deep friction massage and last two weeks electrotherapy and exercise totally 15 session of treatment were applied whi
  Interventions: Other: deep friction massage,; Other: electrotherapy; Other: exercise

INTERVENTIONS:
Other: non -surgical spinal decompression therapy — it is a kind of traction therapy, it has an special traction design which can provide intermittent traction as to herniation levels.
  Arms: combine group; spinal decompression group
Other: deep friction massage, — deep friction massage is a kind of massage targeting deep muscles for decreasing pain and increasing function
  Arms: combine group; exercise group
Other: electrotherapy — electrotherapy is consist of hot pack, ultrasound and TENS. electrotherapy agents were help decreasing pain, increasing metabolism of tissues.
  Arms: combine group; exercise group
Other: exercise — special lumbar stabilization exercises were applied in advanced protocol.
  Arms: combine group; exercise group

SUMMARY:
The aim of this study is to determine the effectiveness of three different treatment methods which consists spinal decompression, deep friction massage and exercise. The patients were separated three groups Group one received non-surgical spinal decompression therapy, group two received non-surgical spinal decompression, lumbar stabilization exercises and manual therapy, group three received manual therapy and lumbar stabilization exercises. All groups completed 15 sessions of therapy. In each session, pain severity was assessed with numeric analog scale, straight leg raise test applied and the degree of the hip flexion where the patient reported pain were recorded, respectively. Static, dynamic muscle strength-endurance tests were applied before the treatment sessions started, after the treatment sessions ended, six weeks after and three months after the study. Oswestry Disability Scale (ODI), Back Performance Scale (BPS), Lanss Neuropathic pain Questionnaire, Fear-Avoidance-Beliefs Questionnaire (FABQ) and McGill Pain Questionnaire were applied before the treatment sessions started, after the treatment sessions ended and three months after the study. Gradient of disc height and thickness of the herniation were assessed segmentally with magnetic resonance imagination (MRI) before the study and three months after the study.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lumbar disc herniation without strengthening loss

Exclusion Criteria:

* clinical diagnosis of osteoporosis
* have scoliosis and spondylolisthesis
* any surgery related spine
* any neurological diseases causes sensory loss

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
magnetic resonance imaging changes | change from baseline in disc height and size of herniation at 3 months.
  changes recorded in micrometrical measurements.

SECONDARY OUTCOMES:
disability | up to 3 months.
  Oswestry Disability Index used to assess the changes in function and disability levels. Scores range from 0 to 100. scores between 0 and 20 described as "minimal disability", scores between 21and 40 described as "moderate disability",scores between 41and 60 described as "severe disability",scores between 61 and 80 described as "crippled" and scores between 81 and 100 described as " bed bounded"
performance | up to 3 months.
  back performance scale used to assess the changes in performance. Scores range from 0 to 15. The lower scores described good performance and higher scores described bad performance.
pain | up to 3 months.
  McGill Pain Questionnaire used to asses the changes in pain levels. scores range from 0 to 78. The higher the pain score the greater the pain.
straight leg raise test for mobility | up to 3 months
  Therapist raised patient's leg passively and the pain felt by the patient measured with goniometer and the angle recorded.
neuropathic pain | up to 3 months.
  The Leeds Assessment of Neuropathic Symptom and Signs (LANSS) Pain Scale used to assess neuropathic pain. Scores range from 0 to 24. scores higher from 12 described neuropathic pain.
fear avoidance beliefs | up to 3 months.
  FABQ used to assess fear related attitudes of the patients. Scores range from 0 to 42 . Higher points described high fear avoidance beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: aynur demirel, PhD, Principal Investigator — Hacettepe University

REFERENCES:
- [Background] Apfel CC, Cakmakkaya OS, Martin W, Richmond C, Macario A, George E, Schaefer M, Pergolizzi JV. Restoration of disk height through non-surgical spinal decompression is associated with decreased discogenic low back pain: a retrospective cohort study. BMC Musculoskelet Disord. 2010 Jul 8;11:155. doi: 10.1186/1471-2474-11-155. PMID 20615252
- [Background] Daniel DM. Non-surgical spinal decompression therapy: does the scientific literature support efficacy claims made in the advertising media? Chiropr Osteopat. 2007 May 18;15:7. doi: 10.1186/1746-1340-15-7. PMID 17511872
- [Background] Lundon K, Bolton K. Structure and function of the lumbar intervertebral disk in health, aging, and pathologic conditions. J Orthop Sports Phys Ther. 2001 Jun;31(6):291-303; discussion 304-6. doi: 10.2519/jospt.2001.31.6.291. PMID 11411624
- [Background] Ozturk B, Gunduz OH, Ozoran K, Bostanoglu S. Effect of continuous lumbar traction on the size of herniated disc material in lumbar disc herniation. Rheumatol Int. 2006 May;26(7):622-6. doi: 10.1007/s00296-005-0035-x. Epub 2005 Oct 25. PMID 16249899
- [Background] Choi J, Lee S, Hwangbo G. Influences of spinal decompression therapy and general traction therapy on the pain, disability, and straight leg raising of patients with intervertebral disc herniation. J Phys Ther Sci. 2015 Feb;27(2):481-3. doi: 10.1589/jpts.27.481. Epub 2015 Feb 17. PMID 25729196
- [Background] Liddle SD, Baxter GD, Gracey JH. Exercise and chronic low back pain: what works? Pain. 2004 Jan;107(1-2):176-90. doi: 10.1016/j.pain.2003.10.017. PMID 14715404
- [Background] Schoenfeld AJ, Weiner BK. Treatment of lumbar disc herniation: Evidence-based practice. Int J Gen Med. 2010 Jul 21;3:209-14. doi: 10.2147/ijgm.s12270. PMID 20689695
- [Background] Meszaros TF, Olson R, Kulig K, Creighton D, Czarnecki E. Effect of 10%, 30%, and 60% body weight traction on the straight leg raise test of symptomatic patients with low back pain. J Orthop Sports Phys Ther. 2000 Oct;30(10):595-601. doi: 10.2519/jospt.2000.30.10.595. PMID 11041196